CLINICAL TRIAL: NCT03371849
Title: A Randomized, Open Label, Single Dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of HCP1102 in Comparison to HGP0813 and HGP1408 Administered in Healthy Male Volunteers
Brief Title: PK and Safety Study of HCP1102, HGP0813 and HGP1408
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HM-MOLZ-103
Record Dates: First submitted 2017-11-24; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — montelukast; levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Reference Drug → Test Drug
  Interventions: Drug: montelukast and levocetirizine FDC; Drug: Singulair + xyzal
- Group 2 (Experimental): Test Drug → Reference Drug
  Interventions: Drug: montelukast and levocetirizine FDC; Drug: Singulair + xyzal

INTERVENTIONS:
Drug: montelukast and levocetirizine FDC — HCP1102
Drug: Singulair + xyzal — HGP0813 + HGP1408

SUMMARY:
This study is a randomized, open label, single dose, two-way crossover clinical trial to investigate the pharmacokinetics and safety/tolerability of HCP1102 in comparison to HGP0813 and HGP1408 administered in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy male volunteers
2. BMI is more than 19kg/m^2 , no more than 28.0 kg/m^2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
AUClast of Montelukast | 1 Day 0 hour, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hour, 2 Day 0 hour, 3 Day 0 hour
Cmax of Montelukast | 1 Day 0 hour, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hour, 2 Day 0 hour, 3 Day 0 hour
AUClast of Levocetirizine | 1 Day 0 hour, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hour, 2 Day 0 hour, 3 Day 0 hour
Cmax of Levocetirizine | 1 Day 0 hour, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 hour, 2 Day 0 hour, 3 Day 0 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moon SJ, Yu KS, Jung J, Kim YI, Kim MG. Comparative pharmacokinetics of a montelukast/levocetirizine fixed-dose combination chewable tablet versus individual administration of montelukast and levocetirizine after a single oral administration in healthy Korean male subjects . Int J Clin Pharmacol Ther. 2020 Jun;58(6):354-362. doi: 10.5414/CP203709. PMID 32271144